CLINICAL TRIAL: NCT03190512
Title: The Effect of Periodontal Treatment on Depression, Body Image, Self-Esteem and Anxiety in Depressed Patients: A Randomized Controlled Clinical Trial
Brief Title: Periodontal Treatment and Psychology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ozge Gokturk (Other)
Responsible Party: Sponsor-Investigator, Ozge Gokturk, Principal Investigator, Tokat Gaziosmanpasa University
Organization: Tokat Gaziosmanpasa University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 14-KAEK-218
Record Dates: First submitted 2017-06-12; First posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Gum Disease
Keywords: Periodontal disease; depression; body image; self-esteem
MeSH Terms: conditions — Gingival Diseases; Periodontal Diseases; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Active Comparator): Psychological measurements were taken from periodontal disease patients before treatment and after 6 weeks.
  Intervention: Non-surgical periodontal treatment (SRP and oral hygiene instructions) was performed and the Psychological questionnaires were filled.
  Interventions: Other: Psychological measurements
- Control Group (Placebo Comparator): Psychological measurements were taken from periodontal disease patients at the baseline and after 6 weeks without the periodontal treatment.
  Intervention: The Psychological questionnaires were filled.
  Interventions: Other: Psychological measurements

INTERVENTIONS:
Other: Psychological measurements — Four questionnaire tests for depression, body image, self-esteem, and anxiety was performed baseline and after 6 weeks.

SUMMARY:
There is a relationship between depression and periodontal disease. This relationship may be double-sided. A psychological state such as anxiety, depression, body image, and self-esteem may be affected from the symptoms of periodontal disease.

DETAILED DESCRIPTION:
Background: Depression is a multi-factorial disease characterized by a variety of symptoms. Psychiatric disorders seem to be more prone to periodontitis compared to patients without psychiatric disorders. However periodontal disease and depression can be considered bidirectional risk factors. Periodontal disease can also be an effect on depression. The aim of this randomized controlled clinical study is to determine the effect of non-surgical mechanical periodontal treatment on psychological state.

Material and methods: The study population consisted of 184 depressed patients with non-treated periodontal diseases. Two randomized group is formed from these patients. Immediately periodontal treatment (test group, n = 92) and delayed periodontal treatment (control group, n = 92). Clinical periodontal and psychological measures were performed at baseline and 6th weeks on control and test group.

ELIGIBILITY:
Inclusion Criteria:

* the presence of periodontal diseases,
* the presence of diagnosed minor depression
* being under maintenance therapy regarding the depression

Exclusion Criteria:

* any hormonal condition such as pregnancy or lactation
* received any periodontal treatment within six months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 184 (Actual)
Dates: Start 2015-05-04 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
Depression level | Baseline and after 6 weeks
  The changes in depression level within 6 weeks. Depression level was determined using the Beck Depression Inventory.

SECONDARY OUTCOMES:
Body image level | Baseline and after 6 weeks
  The changes in body image level within 6 weeks. Body image level was determined using the Body Cathexis Scale.
Anxiety level | Baseline and after 6 weeks
  The changes in anxiety level within 6 weeks. Anxiety level was determined using the Beck Anxiety Inventory.
Self-esteem level | Baseline and after 6 weeks
  The changes in self-esteem level within 6 weeks. Self-esteem level was determined using the Rosenberg Self-Esteem Scale.
Probing pocket depth | Baseline and after 6 weeks
  The changes in probing pocket depth after periodontal treatment.Probing pocket depth was measured for determining severity of disease and clinic outcome.
Clinical attachment level | Baseline and after 6 weeks
  The changes in clinical attachment level after periodontal treatment. Clinical attachment level was measured for determining severity of disease and clinic outcome.
Gingival index | Baseline and after 6 weeks
  The changes in gingival index level after periodontal treatment. Clinical attachment level was measured for determining severity of disease and clinic outcome.
Plaque index | Baseline and after 6 weeks
  The changes in plaque index after periodontal treatment. Plaque index was recorded for determining and classifying oral hygiene status.
Bleeding on probing | Baseline and after 6 weeks
  The changes in bleeding on probing after periodontal treatment. Bleeding on probing was recorded for classifying and evaluating (apically) gingival inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Ozge Gokturk, Principal Investigator — Gaziosmanpasa Universty
Locations (1):
- Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No